CLINICAL TRIAL: NCT06071884
Title: Evaluation of Bridge Device in Pain Management for Outpatient Rotator Cuff Surgery
Brief Title: Bridge Device for Surgical Pain for Rotator Cuff Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Orebaugh (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor-Investigator, Steven Orebaugh, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23030139
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2024-08

CONDITIONS: Pain; Rotator Cuff Injuries
MeSH Terms: conditions — Pain; Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bridge Percutaneous Nerve Field Stimulator (Experimental): The case group (n = 15) will receive an activated Bridge device after surgery and continuing wearing the device until post-operative day (POD) 7.
  Interventions: Device: Bridge Percutaneous Nerve Field Stimulator
- Historical Control (No Intervention): Historical Controls (n=27) who previously had arthroscopic ambulatory rotator cuff surgery, all other factors are the same as the intervention group (multimodal analgesia, etc.)

INTERVENTIONS:
Device: Bridge Percutaneous Nerve Field Stimulator — The Bridge device is an FDA-cleared, drug-free, non-surgical device that uses neuro-modulation to aid in the reduction of symptoms associated with opioid withdrawal through application to branches of the Cranial Nerves V, VII, IX, X, and the occipital nerves. This study is investigating its effectiveness treating post-surgical pain.
  Other Names: NSS-2 BRIDGE
  Arms: Bridge Percutaneous Nerve Field Stimulator

SUMMARY:
The objective of the trial is to investigate the efficacy of the Bridge device in reducing post-operative pain and post-operative opioid consumption in patients undergoing rotator cuff surgery with the typical mode of anesthesia, nerve block plus propofol sedation.

DETAILED DESCRIPTION:
The interscalene block is the gold standard for postoperative pain management following rotator cuff surgery. However, the duration of the block does not cover rehabilitation. Therefore, in most cases, patients are discharged from the surgical center with an opioid prescription. There is a growing need to investigate complementary, non-pharmacologic pain-management methods. The Bridge device, which provides auricular neuromodulation of various cutaneous nerves near the ear, is manufactured by Masimo and previously FDA-approved to reduce symptoms of opioid withdrawal. It is a promising technology that could help relieve post-operative pain without exposing patients to the adverse effects of opioids or other pain-relieving medications. The objective of the trial is to investigate the efficacy of the Bridge device in reducing post-operative pain and post-operative opioid consumption in patients undergoing rotator cuff surgery with the typical mode of anesthesia, nerve block plus propofol sedation. Those enrolled will be assigned to a study group and compared to historic cohort (control group). Historic control group involves patients that underwent same surgical procedure performed at the surgical center involved in the study, by the same surgical operator, between 2020 and 2023.

*Prior to study enrollment, the outcome measure timepoints were updated to postoperative days (POD) 1, 3, 5, and 7. This was largely due to pain trajectories in surgical populations often follow a predictable, nonlinear course, with meaningful fluctuations most apparent on alternating days rather than daily increments. By assessing the outcome measures on POD 1, 3, 5, and 7, the revised scheduled timepoints continues to capture initial peak (POD 1), early recovery phase (POD3), the late recovery phase (POD 5), and the resolution/transition phase (POD 7) regarding pain trajectories.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Willing and able to provide informed consent
* Scheduled to undergo elective rotator cuff surgery at UPMC
* No pre-existing medical conditions which would prevent application of the Bridge device on auricle of ear (i.e., skin infection, rash)

Exclusion Criteria:

* Opioids dependence
* Chronic pain condition with daily opioid use
* Anatomical malformation, which may interfere with placement of the nerve block
* Raynaud's disease diagnosis
* Vasculopathy
* Hemophilia or other coagulopathy, or use of active anticoagulation other than aspirin
* Patient refusal
* Pacemaker
* Pre-existing medical conditions which would prevent application of the Bridge device on auricle of ear (i.e., skin infection, rash)
* Psoriasis vulgaris

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Orebaugh, MD, Principal Investigator — University of Pittsburgh; Amy Monroe, MPH, MBA, Study Director — University of Pittsburgh
Locations (1):
- UPMC Outpatient Center, West Mifflin, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Historical Controls: Historical Controls (n=27) who previously had arthroscopic ambulatory rotator cuff surgery, all other factors are the same as the intervention group (multimodal analgesia)
Period: Overall Study
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Started | 15 | 27
Completed | 15 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population included BRIDGE participants (n = 15) and historical controls (n = 27), for a total of N = 42. Historical controls were identified retrospectively from medical records. Race and ethnicity data were not available for historical controls; therefore, these variables are reported as "Unknown" below.
Groups:
- Historical Controls: Historical Controls (n=27) who previously had arthroscopic ambulatory rotator cuff surgery, all other factors are the same as the intervention group (multimodal analgesia, etc.)
- Total: Total of all reporting groups
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls | Total
Number analyzed (Participants) | 15 | 27 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (6.4) | 56.2 (7.8) | 57.25 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 9 | 15 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity pertaining to historical control group (n=27) unavailable from retrospective medical records review. As a result, ethnicity is reported as "Unknown or Not Reported" below.
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 14 | 0 | 14
    Unknown or Not Reported | 0 | 27 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race pertaining to historical control group (n=27) unavailable from retrospective medical records review. As a result, race is reported as "Unknown or Not Reported" below.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 0 | 0 | 0
    White | 14 | 0 | 14
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 27 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 27 | 42
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.5 (8.1) | 32.3 (7.8) | 31.4 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Oral Opioid Use POD 1
Description: This outcome will be measured by total Oral Morphine Equivalents (OME, mg) abstracted from the medical records.
Time Frame: Post-Operative Day 1
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 27
mg OME | 35.7 (37.1) | 40.2 (28.5)

2. Primary Outcome: Oral Opioid Use POD 3
Description: This outcome will be measured by total Oral Morphine Equivalents (OME, mg) abstracted from the medical records.
Time Frame: Post-Operative Day 3
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 27
mg OME | 21.5 (20.9) | 35.4 (25.7)

3. Primary Outcome: Oral Opioid Use POD 5
Description: This outcome will be measured by total Oral Morphine Equivalents (OME, mg) abstracted from the medical records.
Time Frame: Post-Operative Day 5
Population: Historical Controls data for this outcome were unavailable, and this measure was collected only in the BRIDGE group. Therefore, zero Historical Controls participants were analyzed.
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
mg OME | 6.0 (17.2) |

4. Secondary Outcome: Self-Reported Pain Scores POD 1
Description: Pain scores will be completed on a Numeric Rating Scale (NRS) of 0=no pain at all and 10=the most severe pain.
Time Frame: Post-Operative Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 27
score on a scale | 4.57 (2.9) | 6.42 (2.58)

5. Secondary Outcome: Self-Reported Pain Scores POD 3
Description: Pain scores will be completed on a Numeric Rating Scale (NRS) of 0=no pain at all and 10=the most severe pain.
Time Frame: Post-Operative Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 27
score on a scale | 3.18 (2.2) | 6.75 (2.01)

6. Secondary Outcome: Self-Reported Pain Scores POD 5
Description: Pain scores will be completed on a Numeric Rating Scale (NRS) of 0=no pain at all and 10=the most severe pain.
Time Frame: Post-Operative Day 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
score on a scale | 2.42 (2.1) |

7. Secondary Outcome: Number of Participants Who Self-Reported Oral Opioid Use POD 5
Description: Collected through the subject diary (response yes/no) and recorded as a count of participants
Time Frame: Post-Operative Day 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 7 |
  Responded 'No' | 8 |

8. Secondary Outcome: Number of Participants Who Self-Reported Oral Opioid Use POD 7
Description: Collected through the subject diary (response yes/no) and recorded as a count of participants
Time Frame: Post-Operative Day 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 3 |
  Responded 'No' | 12 |

9. Secondary Outcome: Adverse Events Related to Opioid POD 5
Description: Recorded as yes/no for adverse events related to opioids like nausea, vomiting, dizziness, and itching
Time Frame: Post-Operative Day 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 0 |
  Responded 'No' | 15 |

10. Secondary Outcome: Adverse Events Related to Opioid POD 7
Description: Recorded as yes/no for adverse events related to opioids like nausea, vomiting, dizziness, and itching
Time Frame: Post-Operative Day 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 3 |
  Responded 'No' | 12 |

11. Secondary Outcome: Local Adverse Events on Ear Related to Device POD 1
Description: Recorded as yes/no for adverse events related to the device such as pain or skin irritation
Time Frame: Post-operative Day 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 0 |
  Responded 'No' | 15 |

12. Secondary Outcome: Local Adverse Events on Ear Related to Device POD 3
Description: Recorded as yes/no for adverse events related to the device such as pain or skin irritation
Time Frame: Post-operative Day 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 0 |
  Responded 'No' | 15 |

13. Secondary Outcome: Local Adverse Events on Ear Related to Device POD 5
Description: Recorded as yes/no for adverse events related to the device such as pain or skin irritation
Time Frame: Post-operative Day 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Bridge Percutaneous Nerve Field Stimulator: The case group (n = 15) will receive an activated Bridge device after surgery and continuing wearing the device until post-operative day (POD) 5.
  Bridge Percutaneous Nerve Field Stimulator: The Bridge device is an FDA-cleared, drug-free, non-surgical device that uses neuro-modulation to aid in the reduction of symptoms associated with opioid withdrawal through application to branches of the Cranial Nerves V, VII, IX, X, and the occipital nerves. This study is investigating its effectiveness treating post-surgical pain.
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 0 |
  Responded 'No' | 15 |

14. Secondary Outcome: Local Adverse Events on Ear Related to Device POD 7
Description: Recorded as yes/no for adverse events related to the device such as pain or skin irritation
Time Frame: Post-operative Day 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
Participants
  Responded 'Yes' | 3 |
  Responded 'No' | 12 |

15. Primary Outcome: Oral Opioid Use POD 7
Description: This outcome will be measured by total Oral Morphine Equivalents (OME, mg) abstracted from the medical records.
Time Frame: Post-Operative Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
mg OME | 0.5 (1.94) |

16. Secondary Outcome: Self-Reported Pain Scores POD 7
Description: Pain scores will be completed on a Numeric Rating Scale (NRS) of 0=no pain at all and 10=the most severe pain.
Time Frame: Post-Operative Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
Number analyzed (Participants) | 15 | 0
score on a scale | 1.8 (1.82) |

ADVERSE EVENTS:
Time Frame: 1-week
Description: Adverse events are reported separately for each arm. BRIDGE participants (n=15) were assessed prospectively during the 1-week postoperative period. Historical Controls (n=27) were identified retrospectively, and adverse events were abstracted from available medical records. For outcomes where Historical Controls data were not available, zero Historical Controls participants were analyzed for those outcomes.
Arm/Group | Bridge Percutaneous Nerve Field Stimulator | Historical Controls
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/27
Other Adverse Events (participants affected / at risk) | 3/15 | 5/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bridge Percutaneous Nerve Field Stimulator (N=15) | Historical Controls (N=27)
Skin irritation (Product Issues) | 2 (2) | 0 (0) — Skin irritation related to the device
Continuous electrical stimulation from device (Product Issues) | 1 (1) | 0 (0)
Headache (Surgical and medical procedures) | 0 (0) | 2 (2)
Nausea (Surgical and medical procedures) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT06071884/Prot_SAP_000.pdf